CLINICAL TRIAL: NCT02101060
Title: Effect of Exercise Training on Inflammation and Function in HIV Infected Veterans
Brief Title: Strength Training and Endurance Exercise for LIFE
Acronym: STEEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: O0667-R
Record Dates: First submitted 2014-03-18; First posted 2014-04-01 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: HIV
Keywords: exercise; aging; aerobic capacity; cardiac function; inflammation
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise (Experimental): 16-week progressive aerobic and resistance exercise training
  Interventions: Other: exercise
- control (No Intervention): usual care controls

INTERVENTIONS:
Other: exercise — 16-week progressive aerobic and resistance exercise training
  Arms: exercise

SUMMARY:
Research is needed to determine safe and effective exercise rehabilitation programs to prevent and improve physical disability in older adults living with HIV. This problem is of great importance to the VA. The majority of the 25 thousand HIV-infected veterans are over 50 years of age (64%). The combined effect of aging and inflammation increase the risk for physical disability in older HIV-infected veterans. This translational exercise training trial will examine the cardiac and skeletal muscle effects of combined aerobic exercise and resistance training to attenuate the functional declines of aging with HIV by reducing the deleterious consequences of chronic inflammation. Findings will guide future rehabilitation research on cardiac remodeling and inflammation of skeletal muscle. The proposed research will advance the goal to develop effective rehabilitation strategies that improve the health of older HIV-infected veterans.

DETAILED DESCRIPTION:
The objective of this study is to determine the effect of exercise training on the central (cardiovascular) and peripheral (muscular) impairments underlying poor physical function by comparing older HIV-infected veterans randomized to combine aerobic and resistance exercise training versus usual care. The study hypothesis is that a progressive aerobic and resistance rehabilitation program will increase aerobic capacity and muscle strength, which will be mediated by improved diastolic function, increased muscle mass, and decreased systemic inflammation. To test this hypothesis, investigators will conduct a randomized 16-week trial of progressive aerobic and resistance training versus usual care control in 40 sedentary older (50+ years) HIV-infected veterans. The study will determine the effects of exercise training on aerobic capacity and diastolic function, and their relationship to changes in biomarkers of systemic inflammation and cardiac fibrosis (AIM 1). The study will also determine the effect of exercise training on strength and muscle mass, and their relationship to changes in biomarkers of systemic inflammation (AIM 2).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected veterans adult 50 years of age and older under medical care for HIV
* Antiretroviral Therapy

Exclusion Criteria:

* Patients with comorbid conditions that could have a potential impact on their ability to perform exercise testing and training will be excluded according to the American College of Sports Medicine
* Only sedentary adults will be eligible. Individuals that participate in regular structured aerobic exercise or resistance training in the prior 6-months will be excluded

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann K Oursler, MD, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Salem VA Medical Center, Salem, VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Briggs BC, Ryan AS, Sorkin JD, Oursler KK. Feasibility and effects of high-intensity interval training in older adults living with HIV. J Sports Sci. 2021 Feb;39(3):304-311. doi: 10.1080/02640414.2020.1818949. Epub 2020 Sep 23. PMID 32962523
- [Result] Oursler KK, O'Boyle HM, Briggs BC, Sorkin JD, Jarmukli N, Katzel LI, Freiberg MS, Ryan AS. Association of Diastolic Dysfunction with Reduced Cardiorespiratory Fitness in Adults Living with HIV. AIDS Patient Care STDS. 2019 Dec;33(12):493-499. doi: 10.1089/apc.2019.0149. PMID 31821043
- [Result] Oursler KK, Iranmanesh A, Jain C, Birkett KL, Briggs BC, Garner DC, Sorkin JD, Ryan AS. Short Communication: Low Muscle Mass Is Associated with Osteoporosis in Older Adults Living with HIV. AIDS Res Hum Retroviruses. 2020 Apr;36(4):300-302. doi: 10.1089/AID.2019.0207. Epub 2019 Dec 23. PMID 31762303
- [Result] Ryan AS, Roy A, Oursler KK. Gait and Balance Biomechanics in Older Adults With and Without Human Immunodeficiency Virus. AIDS Res Hum Retroviruses. 2019 Nov/Dec;35(11-12):1089-1094. doi: 10.1089/AID.2019.0102. PMID 31547668

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | Control
Started | 17 | 16
Completed | 12 | 12
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Control | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.03 (6.1) | 61.17 (7.4) | 61.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 9 | 23
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Aerobic Capacity
Description: VO2 peak will be used as the primary measure of aerobic capacity. Subjects will be asked to exercise to voluntary exhaustion during a treadmill test using a modified Bruce protocol.
  In this Outcome, a mean difference between baseline to 16 weeks is reported (value at 16 weeks minus value at baseline).
Time Frame: at baseline and at 16 weeks (before and after the intervention phase)
Population: We have incomplete data on completers in the control group.
Measure: Mean (Standard Error); unit: Liters/minute
Arm/Group | Exercise | Control
Number analyzed (Participants) | 12 | 11
Liters/minute | 0.15 (0.04) | 0.02 (0.07)

2. Primary Outcome: Diastolic Function
Description: Exercise stress two-dimensional transthoracic echocardiography with tissue Doppler imaging (stress-echo) will be used to collect data on diastolic function. Reporting on ejection fraction.
  In this Outcome, a mean difference between baseline to 16 weeks is reported (value at 16 weeks minus value at baseline).
Time Frame: at baseline and at 16 weeks (before and after the intervention phase)
Population: We have incomplete data on completers in these groups.
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Exercise | Control
Number analyzed (Participants) | 11 | 10
percentage | 1.8 (1.9) | 0.5 (2.7)

3. Secondary Outcome: Biomarkers of Systemic Inflammation
Description: Changes in plasma levels of biomarkers of chronic inflammation will be calculated pre/post intervention, and will be tested for association with changes in primary outcomes as well as between group differences. Presenting IL-18 values (log converted for analysis).
  In this Outcome, a mean difference between baseline to 16 weeks is reported (value at 16 weeks minus value at baseline).
Time Frame: at baseline and at 16 weeks (before and after the intervention phase)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Exercise | Control
Number analyzed (Participants) | 12 | 12
pg/mL | -0.04 (0.02) | -0.03 (0.02)

ADVERSE EVENTS:
Time Frame: Data collected from time of enrollment to completion of study. For intervention group, duration of study is approximately 30 weeks. For control group, duration of study is approximately 50 weeks.
Arm/Group | Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=17) | Control (N=16)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — reoccurrence of pre-existing Supraventricular tachycardia
dizziness (Cardiac disorders) | 0 (0) | 1 (1) — In delayed entry exercise of control group
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — In delayed entry exercise of control group

LIMITATIONS AND CAVEATS:
Exclusion criteria may limit the generalizability of findings. While AIDS-related conditions are an exclusion criteria, the period is limited to the prior 6 months. In order to minimize confounding by ART medication, we require participants to be on the same regimen for at least 3 months prior to enrollment. Therefore, we have included a control group without exercise and assume that the risk of confounding from ART and other medications will be equally distributed across groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02101060/Prot_SAP_000.pdf